CLINICAL TRIAL: NCT01124526
Title: Prospective Non-randomized Multicenter Study to Assess the Efficacy Response Duration and Toxicity of RFC as First-line Treatment and R as Maintenance Treatment, in Patients Diagnosed of Follicular Non Hodgkin Lymphoma
Brief Title: Efficacy Response Duration and Toxicity of Rituximab, Fludarabine, and Cyclophosphamide (RFC) as 1st Line Treatment and Rituximab (R) in Maintenance Treatment in Follicular Non Hodgkin (FNH) Lymphoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asociacion Espanola de Hematologia y Hemoterapia (Other)
Responsible Party: JF Tomás / MD, Asociación Española de Hematología y Hemoterapia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNHF-03.; 04-0199 (Other: Spanish Health Minyster (AEMPS)); 2004/254 (Other: Local Ethic Comities from Madrid CEIC_R MADRID)
Record Dates: First submitted 2009-02-10; First posted 2010-05-17 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Non Hodgkin Lymphoma
Keywords: R F C treatment in patients with Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab, Fludarabine, ciclophosphamide (Experimental): Patients receiving from 4 to 6 cycles of chemotherapy (R F C) each 4 weeks depending on haematological tolerance:
  RITUXIMAB(R)375 mg/m2 iv,day 3 C1 and day 1 C2-C6,(total dose 375 mg/m2)
  Interventions: Drug: Rituximab Fludarabine Cyclophosphamide

INTERVENTIONS:
Drug: Rituximab Fludarabine Cyclophosphamide — Patients receiving from 4 to 6 cycles of chemotherapy (R F C) each 4 weeks depending on haematological tolerance:
  RITUXIMAB(R)375 mg/m2 iv,day 3 C1 and day 1 C2-C6,(total dose 375 mg/m2) FLUDARABINE(F):25 mg/m2 iv, day 1-3,(total dose 75 mg/m2) CICLOPHOSPHAMIDE(C)1000 mg/m2 iv, day 1,(total dose 1000 mg/m2)
  Other Names: MABTHERA; BENEFLUR; GENOXAL

SUMMARY:
The purpose of this study is to determine whether the rituximab administration with fludarabine and cyclophosphamide results, are better, than the ones obtained with conventional therapy such as CHOP (cyclophosphamide, adriamycin, vincristine, prednisone) and also to determine whether the rituximab administration as maintenance treatment during two years, increase the global clinical responses and the disease free time interval.

DETAILED DESCRIPTION:
The use of monoclonal antibodies, specifically the chimerical humanized anti-CD20 monoclonal antibody (Rituximab, MabThera®) represents one of the most innovative aspects in the indolent lymphoma treatment. Preliminary data show from 40% to 50% of response with a median response duration between 6 and 11 months in patients with relapsing FL. This response rate increase when rituximab is administered as initial treatment.

Therefore, not only due to the clinical results but also to the tolerance, and based on an innovative mechanism of action and in its minimal toxicity, it seems reasonable to raise the possibility to incorporate the administration of the monoclonal antibody with chemotherapeutic agents.

The development of a new treatment scheme that includes Rituximab administration within treatment protocols that combine fludarabine and cyclophosphamide, whose results are better than the ones obtained with conventional treatments such as CHOP, should increase the molecular response rate and contribute therefore to increase the disease-free time interval (time to progression), without adding any toxicity, in addition to achieve a higher proportion of clinical responses (as global as complete responses). In order to increase the time interval to progression, a maintenance treatment will be carried out for 2 years, which has shown an evident benefit in the time to progression in preliminary studies.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with grade I-III follicular lymphoma (grade B- D from the Working Formulation, centrofollicular lymphoma in the REAL classification), without evidence of histological transformation.
* Clinical diagnose by histological and/or immunophenotypical evaluation with positive results for CD 20 Mo Ab (node, bone marrow).
* Ann-Arbor stage II-IV.
* Male and female patients from 18 to 75 years old.
* Lack of related clinically uncontrolled diseases.
* Lack of VIH infection.
* Performance status (ECOG) of 0, 1, 2.
* Patients who voluntarily gave informed consent for the study participation.
* Life expectancy > 3 months.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Women of childbearing age who do not accept to use an effective contraceptive method during the treatment and one year post-treatment.
* Immunodeficiency condition and autoimmune diseases.
* Patients with advanced clinically uncontrolled cardiac, hepatic or renal insufficiency, defined by the following criteria: total bilirubin, alkaline phosphatase or transaminases >2 x upper limit of normal, and serum creatinine value >2 x upper limit of normal.
* Patients previously treated with chemotherapy or radiotherapy.
* History of oncologic disease within the last 5 years, apart from non-melanoma cutaneous neoplasia or carcinoma in situ of uterine cervix.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2004-09; Primary Completion 2007-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Time to progression disease | 42 months

SECONDARY OUTCOMES:
Free-disease period | 54 months
Overall survival | 54 months
Safety of RFC | 54 months
  Toxicity is detailed and tabulate following the WHO classification. The safety analysis includes the incidence of adverse events (AE),vital signs and laboratory parameters.
  Impact tables are made of AE following the classification of preferred term. Also include an analysis of the intensity of AE and their relation to the combiantion of study treatment.
Molecular monitoring of clinical response | 54 months
  Study of t14:18 translocation with altered expression of BCL2.

CONTACTS AND LOCATIONS:
Overall Officials: José F. Tomás, MD, Study Director — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; E . Prieto Pareja, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; F. Hernández Navarro, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; J. Díaz Mediavilla, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; C. Montalbán, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; F. Javier Peñañver, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; J. De La Serna, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; Mª Carmen Burgaleta, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; P. Sánchez Godoy, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; Mª Dolores Monteagudo, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; A. Fernández De Sevilla, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; Mª Jesús Peñarrubia, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; Mª Dolores Caballero Barrigón, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; R. Bajo Gómez, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; A. Paz Coll, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; J. A. Queizán, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; C. Cabrera Silva, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; O. Arija, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; P. Bravo Barahona, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon; A. Salar, MD, Principal Investigator — Fundacion para el Estudio de la Hematologia y Hemoterapia en Aragon
Locations (20):
- Spain (20):
  - Hospital Infanta Cristina, Badajoz, Badajoz_Extremadura
  - Hospital del Mar, Barcelona, Barcelona_ Cataluña
  - Instituto Catalán de Oncología (ICO), Barcelona, Barcelona_Cataluña
  - Hospital San Pedro de Alcántara, Cáceres, Cáceres_Extremadura
  - Hospital de Puerto Real, Puerto Real, Cádiz_ Andalucía
  - Complejo Hospitalario Xeral_Calde, Lugo, Lugo_ Galicia
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Fundación Hospital Alcorcón, Alcorcón, Madrid
  - Hospital de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Severo Ochoa, Leganés, Madrid
  - MD Anderson Internacional España, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital de Móstoles, Móstoles, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca, Salamanca_Castilla León
  - Hospital General de Segovia, Segovia, Segovia_ Castilla León
  - Hospital Clínico del Río Hortega, Valladolid, Valladolid_Castilla León